CLINICAL TRIAL: NCT05411263
Title: Portal Vein Flow Variability to Quantify Right-Sided Hemodynamic Congestion: A Proof-Of-Concept Study
Brief Title: Portal Vein Flow Variability to Quantify Right-Sided Hemodynamic Congestion (PORTAL)
Acronym: PORTAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: HeartKinetics (Unknown)
Responsible Party: Principal Investigator, Frederik Hendrik Verbrugge, MD PhD MSc, Clinical Professor/Head of Clinic, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC-2021-268
Record Dates: First submitted 2022-05-31; First posted 2022-06-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Congestion; Heart Failure; Right Heart Catheterisation; Central Venous Pressure; Doppler Echocardiography
Keywords: Congestion; Doppler echocardiography; Central venous pressure; Right heart catheterisation; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced heart failure undergoing clinically indicated right heart catheterisation (Experimental): Patients with advanced heart failure undergoing right heart catheterisation as clinically indicated, irrespectively of their ejection fraction.
  Interventions: Diagnostic Test: Comprehensive transthoracic echocardiography, Doppler echography & Kino-cardiograph (Kino)

INTERVENTIONS:
Diagnostic Test: Comprehensive transthoracic echocardiography, Doppler echography & Kino-cardiograph (Kino) — As per inclusion criteria, all patients undergo right heart catheterisation to obtain a full profile of invasive hemodynamic measurements, including pulmonary arterial wedge pressure (PAWP), pulmonary artery pressure, right ventricular pressure, right atrial pressure (RAP), superior and/or inferior vena cava pressure, hepatic vein pressure with/without balloon occlusion. Immediately after the invasive hemodynamic exam, a comprehensive 2D, Color Doppler and Doppler echocardiography exam, including a Doppler study of the Vv. hepaticae, V. portae and V. renalis is performed. Based upon logistic feasibility, ballistocardiography and seismocardiography with the completely non-invasive Kino device (HeartKinetics, Waterloo, Belgium) is performed in a subpopulation of patients envisioned to be at least 50 patients.

SUMMARY:
This study evaluates the accuracy of a comprehensive venous Doppler echography including the portal vein pulsatility index (PVPI) to quantify invasively measured right-sided venous pressures. A substudy will correlate invasive and non-invasive hemodynamic measurements to ballistocardiography and seismocardiography with the Kino-cardiograph (Kino) device (HeartKinetics, Waterloo, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 year old and able to provide informed consent;
* Consecutive patients scheduled for right heart catheterisation by a dedicated heart failure specialist at the Centre of Cardiovascular Diseases (University Hospital Brussels, Jette, Belgium).

Exclusion Criteria:

* Major anatomical variations of the portal veins (agenesis of left and right portal vein) and/or arterio-portal vein fistula;
* Patients with Child-Pugh B or C liver cirrhosis or liver transplant;
* Body Mass Index < 20 kg/m².

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Portal Vein Pulsatility Index (PVPI) | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  PVPI = (Vmax - Vmin)/Vmax on the portal vein Pulsed wave Doppler signal

SECONDARY OUTCOMES:
Time integral of kinetic energy during the cardiac cycle | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  Measured by a combination of ballistocardiography and seismocardiography with the Kino device (HeartKinetics, Waterloo, Belgium).
Inferior vena cava diameter | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  Inferior vena cava diameter [mm] upon end-expiration
Inferior vena cava diameter respiratory variation | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  Inferior vena cava diameter respiratory variation [%]
Hepatic vein Pulsed wave Doppler signal | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  Categorical classification:
  * Systolic wave > Diastolic wave
  * Diastolic wave > Systolic wave
  * Systolic flow reversal
Renal vein Pulsed wave Doppler signal | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  Categorical classification:
  * Monophasic flow
  * Discontinuous biphasic flow
  * Discontinuous monophasic flow
Right ventricular (RV) free wall strain | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  Right ventricular (RV) free wall strain assessed in the RV focused view offline with EchoPAC (General Electric Healthcare, Chicago, IL, United States).
Right atrial strain | Crosssectional study without longitudinal follow-up, measurement is obtained during Doppler echography exam
  Right atrial strain assessed in the RV focused view offline with EchoPAC (General Electric Healthcare, Chicago, IL, United States).

CONTACTS AND LOCATIONS:
Overall Officials: Frederik H Verbrugge, MD; PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- University Hospital Brussels, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data related will be made available upon reasonable request in adherence with transparency conventions in medical research, always through requests addressed to the primary investigator.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year after completion of the study

DOCUMENTS (1):
  • Study Protocol (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT05411263/Prot_000.pdf